CLINICAL TRIAL: NCT00573872
Title: A Phase II Study of Spinal Radiosurgery
Acronym: RAD0408
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: Health Services Foundation (Unknown); The Kirklin Clinic at Acton Road (Unknown)
Responsible Party: Principal Investigator, John Fiveash, MD, Professor and Vice Chair, University of Alabama at Birmingham Department of Radiation Oncology, University of Alabama at Birmingham
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: F050103003; T0408240012
Record Dates: First submitted 2007-12-12; First posted 2007-12-14 (Estimated); Results first posted 2017-10-20 (Actual); Last update posted 2017-12-05 (Actual); Status verified 2017-10

CONDITIONS: Neoplasm; Arteriovenous Malformations
Keywords: Radiosurgery; Phase II; Cancer; Spinal; AVM
MeSH Terms: conditions — Neoplasms; Arteriovenous Malformations | interventions — Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Spinal Radiosurgery (Experimental): Patients will be fitted in a custom immobilization device. A CT simulation scan will then be performed to pinpoint intended radiosurgery target producing a computer optimized radiation plan to be confirmed by planning radiation physicist. Patient will then be placed in their immobilization device and aligned with the treatment planning position. Patient then receives radiosurgery. Treatment delivery will be divided into components of 3-5Gy with repeat CT based localization in between each of these components. For all patients, a nominal prescription dose of 24Gy will be entered into the tomotherapy cost function. Once the plan that provides maximal spinal sparing has been generated, the plan will be renormalized to produce no more than 8Gy (prior RT) or 10Gy (no prior RT) to 0.5cc of spinal cord by dividing the single fraction treatment into fractions of 3-5Gy.
  Interventions: Radiation: Radiosurgery

INTERVENTIONS:
Radiation: Radiosurgery — Phase I: 20-25 Gy in 5 fractions
  Phase II: 9-24 GY in 1 fraction

SUMMARY:
Phase I of the study (motion and quality assurance [QA] study) is being used to determine intrafraction target motion and define quality assurance procedures for single fraction spinal radiosurgery. The Phase II portion of the study is being used to estimate the palliative response (pain or relief of neurologic symptoms) and local control for single fraction radiosurgery delivered with TomoTherapy and to assess the acute and late toxicity of spinal radiosurgery.

DETAILED DESCRIPTION:
Optimal radiation plan is generated that treats the tumor (CTV) and spares normal tissue, especially the spinal cord. Motion and QA study will determine intrafraction motion for phase II portion of the study.

Dose prescription to tumor is based upon maximal dose received by 0.5 cc of spinal cord and whether patient has had prior radiation therapy to that area:

Phase I - Motion and QA Study: 20-25 Gy in 5 fractions/10-20 patients/previous RT = <50% CTV dose/No previous RT = <80% CTV dose.

Phase II - 9-24 Gy in 1 fraction/30 total in order to have 20 evaluable patients (15 patients with prior RT and 15 without prior RT/previous RT = 8 Gy/No previous RT = 10 Gy.

# Motion and QA study will treat CTV to 20-25 Gy in 5 fractions to study intrafraction motion for QA of single fraction administration. This will define treatment margins for single fraction radiosurgery.

*Previous RT:

* greater than six months since completion of RT
* at least 20 Gy, but no more than 50 Gy

ELIGIBILITY:
Inclusion Criteria:

1. All subjects must have history of histologically confirmed neoplasm or radiographically-diagnosed AVM. Patients without a prior tissue diagnosis but who have a radiographically characteristic lesion are eligible if there is consensus agreement of the diagnosis in the UAB Neuro-oncology Tumor Board.
2. ECOG performance status of less than or equal to 2
3. Age greater than 18
4. Life expectancy greater than 12 weeks
5. Subjects given written informed consent

Exclusion Criteria:

1. Cytotoxic chemotherapy within 7 days of treatment
2. Insufficient recovery from all active toxicities of prior therapies
3. Epidural spinal cord compression requiring immediate neurosurgical decompression. If a patient requires immediate surgery for neurologic compromise, they may still be eligible post operatively if tumor was incompletely resected.
4. Patient is non-ambulatory. Optimization of pretreatment neurologic function with steroids is allowed. Ambulation with assistance of walker or cane is allowed.
5. Patient is pregnant and it is judged by the treating Radiation Oncologist that spinal radiosurgery would place the fetus in unacceptable danger.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2005-04 (Actual); Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John B. Fiveash, M.D., Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham/The Kirklin Clinic at Acton Road, Birmingham, Alabama, United States

REFERENCES:
- [Background] Abbatucci JS, Delozier T, Quint R, Roussel A, Brune D. Radiation myelopathy of the cervical spinal cord: time, dose and volume factors. Int J Radiat Oncol Biol Phys. 1978 Mar-Apr;4(3-4):239-48. doi: 10.1016/0360-3016(78)90144-x. No abstract available. PMID 640895
- [Background] Ang KK, Jiang GL, Feng Y, Stephens LC, Tucker SL, Price RE. Extent and kinetics of recovery of occult spinal cord injury. Int J Radiat Oncol Biol Phys. 2001 Jul 15;50(4):1013-20. doi: 10.1016/s0360-3016(01)01599-1. PMID 11429229
- [Background] Bilsky MH, Yamada Y, Yenice KM, Lovelock M, Hunt M, Gutin PH, Leibel SA. Intensity-modulated stereotactic radiotherapy of paraspinal tumors: a preliminary report. Neurosurgery. 2004 Apr;54(4):823-30; discussion 830-1. doi: 10.1227/01.neu.0000114263.01917.1e. PMID 15046647
- [Background] Daut RL, Cleeland CS, Flanery RC. Development of the Wisconsin Brief Pain Questionnaire to assess pain in cancer and other diseases. Pain. 1983 Oct;17(2):197-210. doi: 10.1016/0304-3959(83)90143-4. PMID 6646795
- [Background] Delattre JY, Rosenblum MK, Thaler HT, Mandell L, Shapiro WR, Posner JB. A model of radiation myelopathy in the rat. Pathology, regional capillary permeability changes and treatment with dexamethasone. Brain. 1988 Dec;111 ( Pt 6):1319-36. doi: 10.1093/brain/111.6.1319. PMID 3208060
- [Background] Gerszten PC, Ozhasoglu C, Burton SA, Vogel WJ, Atkins BA, Kalnicki S, Welch WC. CyberKnife frameless stereotactic radiosurgery for spinal lesions: clinical experience in 125 cases. Neurosurgery. 2004 Jul;55(1):89-98; discussion 98-9. PMID 15214977
- [Background] Glanzmann C, Aberle HG, Horst W. The risk of chronic progressive radiation myelopathy. Strahlentherapie. 1976 Oct;152(4):363-72. PMID 982487
- [Background] Nieder C: Recommendation of Human Spinal Cord Re-irradiation Dose Based on Data From 39 Patients. Int J Radiat Oncol Biol Phys 57:373, 2003
- [Background] Schultheiss TE, Stephens LC. Invited review: permanent radiation myelopathy. Br J Radiol. 1992 Sep;65(777):737-53. doi: 10.1259/0007-1285-65-777-737. No abstract available. PMID 1393407
- [Background] Schultheiss TE, Stephens LC, Jiang GL, Ang KK, Peters LJ. Radiation myelopathy in primates treated with conventional fractionation. Int J Radiat Oncol Biol Phys. 1990 Oct;19(4):935-40. doi: 10.1016/0360-3016(90)90015-c. PMID 2211262
- [Background] Schultheiss TE, Stephens LC, Maor MH. Analysis of the histopathology of radiation myelopathy. Int J Radiat Oncol Biol Phys. 1988 Jan;14(1):27-32. doi: 10.1016/0360-3016(88)90046-6. PMID 3275603

RESULTS

PARTICIPANT FLOW:
Groups:
- Spinal Radiosurgery: Patients will be fitted in a custom immobilization device. A CT simulation scan will then be performed to pinpoint intended radiosurgery target producing a computer optimized radiation plan to be confirmed by planning radiation physicist. Patient will then be placed in their immobilization device and aligned with the treatment planning position. Patient then receives radiosurgery. Treatment delivery will be divided into components of 3-5Gy with repeat CT based localization in between each of these components. For all patients, a nominal prescription dose of 24Gy will be entered into the tomotherapy cost function. Once the plan that provides maximal spinal sparing has been generated, the plan will be renormalized to produce no more than 8Gy (prior RT) or 10Gy (no prior RT) to 0.5cc of spinal cord by dividing the single fraction treatment into fractions of 3-5Gy.
  Radiosurgery: Phase I: 20-25 Gy in 5 fractions
  Phase II: 9-24 GY in 1 fraction
Period: Overall Study
Arm/Group | Spinal Radiosurgery
Started | 43 (# of patients that signed consent)
Completed | 32 (# of patients that completed treatment)
Not Completed | 11

BASELINE CHARACTERISTICS:
Arm/Group | Spinal Radiosurgery
Number analyzed (Participants) | 32
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 19
  >=65 years | 13
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 19
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 28
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Palliative Response (Pain or Relief of Neurologic Symptoms) From Single Fraction Radiosurgery Delivered With Tomotherapy
Description: Physician's subjective report of palliative pain relief. The maximal benefit patient received (best response) is reported. Scale is pain described as "worse", "stable", "better", or "completely resolved". In the reporting "better" or "completely resolved" indicates response to treatment.
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Spinal Radiosurgery
Number analyzed (Participants) | 32
Participants | 29

2. Primary Outcome: Assess the Acute and Late Toxicity of Spinal Radiosurgery
Description: CTCAE version 3. Acute toxicity will be recorded if toxicity occurs early phase or within 3 months, and late toxicity would be any toxicity that follows those 3 months.
Time Frame: 2 years
Measure: Number; unit: events
Arm/Group | Spinal Radiosurgery
Number analyzed (Participants) | 43
events | 4

3. Primary Outcome: Number of Participants With Lack of Tumor Growth at Last Follow-up
Description: Lack of tumor growth by CT or MRI at last follow-up
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Spinal Radiosurgery
Number analyzed (Participants) | 32
Participants | 21

ADVERSE EVENTS:
Arm/Group | Spinal Radiosurgery
Serious Adverse Events (participants affected / at risk) | 1/32
Other Adverse Events (participants affected / at risk) | 1/32
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Spinal Radiosurgery (N=32)
Hospitalization for Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Pre protocol treatment, the patient was admitted to hospital for pneumonia. The patient received IV antibiotics and was discharged 3/21/06 on home antibiotics after resolution of pneumonia. The patient was able to receive treatment same day.
Worsening neurological symptoms from progressive spinal disease (Nervous system disorders) | 1 (1) — Over 4 weeks, the patient experienced worsening of neurological symptoms and decreased ability to ambulate. MRI found to have progressive spinal disease. Surgery of the spinal disease revealed metastatic renal cell carcinoma.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Spinal Radiosurgery (N=32)
Grade 2 myelopathy (Nervous system disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No